CLINICAL TRIAL: NCT07222787
Title: Post-market Safety and Effectiveness of the CORUS-LX System in Improving Lumbar Interbody Fusion Outcomes for the Treatment of Degenerative Lumbosacral Disc Disease.
Brief Title: Post-market Safety and Effectiveness of the CORUS-LX System in Improving Lumbar Interbody Fusion Outcomes (ILIF)
Acronym: ILIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMT0004
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Radiculopathy Lumbar; Degenerative Lumbar Disc Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to their assignment through the day of surgery, however will be informed of what treatment they received once the surgery is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Supplemental Posterior Fusion Technique (Active Comparator): Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with standard supplemental posterior fusion including pedicle screw and rod fixation.
  Interventions: Device: Supplemental Posterior Fusion with Standard Technique
- Supplemental Posterior Fusion with Study Device (Experimental): Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with supplemental posterior fusion performed using the study device, including pedicle screw and rod fixation.
  Interventions: Device: Supplemental Posterior Fusion with Study Device

INTERVENTIONS:
Device: Supplemental Posterior Fusion with Study Device — Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with supplemental posterior fusion performed using the Study Device, including pedicle screw and rod fixation.
  Arms: Supplemental Posterior Fusion with Study Device
Device: Supplemental Posterior Fusion with Standard Technique — Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with standard minimally invasive supplemental posterior fusion including pedicle screw and rod fixation.
  Arms: Standard Supplemental Posterior Fusion Technique

SUMMARY:
The goal of this clinical trial is to assess the safety and effectiveness of the study device, CORUS-LX, as an adjunct to lumbar interbody fusion, when used in combination with pedicle screw and rod constructs for the treatment of lumbosacral degenerative disease in patients requiring 2 level (L4-S1) lumbar fusion, for the treatment of symptomatic degenerative lumbosacral disc disease. The main questions it aims to answer are:

Is there fusion success at the treated posterior anatomy of each level? Is there an absence of major adverse device related events? Is there an absence of injections (steroid, facet joint, nerve block) or subsequent revision surgery at index levels for symptoms related to back or leg pain?

Researchers will compare a control arm to the treatment arm to see if research results vary from standard minimally invasive supplemental posterior fusion.

Eligible participants will undergo one of the below interventions:

* Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with supplemental posterior fusion performed using the study device, including pedicle screw and rod fixation.
* Two-level lumbar interbody fusion at L4-L5 & L5-S1 segments, with standard minimally invasive supplemental posterior fusion including pedicle screw and rod fixation.

Participants will also be asked to read, understand, and sign the informed consent, attend a Screening/Baseline visit, undergo surgery for their designated intervention, and participate in 5 additional study visits where they will complete surveys for patient reported outcomes and SOC procedures. These visits will occur at the below intervals (based upon surgery day as day 0):

* 6 weeks
* 3 months
* 6 months
* 12 months
* 24 months

DETAILED DESCRIPTION:
The study device is designed to provide surgeons a tissue-sparing solution for both preparing a fusion bed around the facet space in addition to stabilizing the joint in sync with percutaneous pedicle screw and rod fixation. There have been few rigorous studies looking at the posterior fusion aspect of circumferential lumbar fusion. Through a randomized controlled trial design and multi-modal imaging protocol, we aim to explore whether the opportunity for improved outcomes exists.

This randomized controlled trial was designed to compare outcomes in subjects treated with interbody fusion including supplemental posterior fusion for the treatment of degenerative lumbosacral disease. For the control arm subjects, supplemental posterior fusion will be performed with each surgeon's standard protocol for fusion with pedicle screw and rods. Treatment arm subjects will also receive percutaneous pedicle screw fixation but will also have the posterior anatomy prepared for fusion using the study device. In both arms, all posterior instrumentation will be placed using navigation technology. Study success will be defined as the demonstration of statistical superiority by the treatment arm over the control arm with respect to the primary endpoint, which is the incidence of arthrodesis achieved across the posterior anatomy. Additional data of interest will be collected to explore relationships between observed arthrodesis rates at the posterior anatomy and the rates of arthrodesis across the interbody space, serious device-related adverse events, device failure, subsequent surgical revisions, patient-reported outcomes, and return-to-work measures assessed through 24 months. Eligible subjects will be those with degenerative lumbosacral disease diagnosed at 2 levels between the L4 and S1 segments who are indicated for treatment using an interbody fusion approach supplemented with posterior fusion including pedicle screw and rod fixation. Major exclusionary factors will be history of prior instrumentation at the index or adjacent levels, fused facet or facet hypertrophy that prohibits device implantation, and a diagnosis of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years (Skeletally Mature)
2. Indicated for lumbar interbody fusion for treatment of degenerative lumbosacral disease at two contiguous disc levels between L4-S1 as determined by the following:

   a) Diagnosis of radiculopathy of the lumbar spine, with pain, including at least one of the following: i) Leg and/or buttock pain, weakness, numbness, or paresthesia ii) Low back pain iii) Neurogenic claudication b) Radiographically determined pathology (CT, MRI, X-rays) at the levels to be treated correlating to primary symptoms including at least one of the following: i) Decreased disc height in comparison to a normal adjacent disc. ii) Degenerative instability ≤ grade 1 spondylolisthesis (<25% slip). iii) Recurrent disc herniation. iv) Central and/or foraminal stenosis.
3. Oswestry Disability Index Score of > 40/100 (Severe Disability).
4. Unresponsive to non-operative, conservative treatment (rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics) for:

   1. At least six weeks from symptom onset; or
   2. Have the presence of progressive symptoms or signs of nerve root/ spinal cord compression despite continued non-operative conservative treatment.
5. Reported to be medically cleared for surgery.
6. Physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms
7. Willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.
8. Written informed consent provided by subject.

Exclusion Criteria:

1. Any disease or condition that, in the investigator's opinion, would preclude accurate radiographic evaluation of any treated vertebrae (e.g. morbid obesity).
2. Any anatomy or condition that makes posterior fusion treatment infeasible (e.g. fused facets).
3. Has, in the Investigator's opinion, any disease or condition that would preclude accurate clinical evaluation (e.g. neuromuscular disorders).
4. Active systemic infection or infection at the operative site.
5. Anticipated treatment for active systemic infection, including HIV or Hepatitis C.
6. Previous trauma to any of the L3 to S1 levels resulting in significant bony or disco-ligamentous lumbar spine injury that may prevent device placements.
7. Prior instrumented surgery or pseudoarthrosis at the operative or adjacent levels.
8. Indicated for or history of laminectomy at any of the index or adjacent levels
9. Fixed or permanent neurologic deficit related to the target treatment levels that cannot be improved with surgery
10. Leg, buttocks, or back pain in the absence of other symptoms of radiculopathy or myeloradiculopathy justifying the need for surgical intervention.
11. Symptomatic disc degeneration requiring surgical intervention at more or less than two levels.
12. Diagnosis of spondylolisthesis, grade >1.
13. Diagnosis of lytic spondylolisthesis
14. Diagnosis of iatrogenic, traumatic, or dysplastic spondylolisthesis
15. Congenital bony and/or spinal cord abnormalities affecting spinal stability.
16. Diagnosis of Paget's disease, osteomalacia or any other metabolic bone disease other than osteopenia.
17. Diagnosis of osteoporosis, defined as a previous DEXA bone density T-score of ≤-2.5.
18. Active malignancy or a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and without clinical signs or symptoms of the malignancy for at least five years.
19. Has an uncontrolled seizure disorder.
20. Cauda equina syndrome or neurogenic bowel/bladder dysfunction;
21. Use of epidural steroids within 14 days prior to surgery.
22. A concomitant condition requiring daily, high-dose oral steroids.

    High dose steroid use is defined as:
    1. Daily, chronic use of oral steroids of 5 mg/day or greater (steroid inhalers are not exclusionary).
    2. Use of short-term (less than 10 days) oral steroids at a daily dose greater than 40 mg within one month of the study procedure.
23. Long-term use (>6 months) of opioids >120 mg morphine equivalents.
24. Known allergy to titanium (Ti)
25. A current or recent history (≤1 year prior to screening) of substance abuse that required medical treatment.
26. Is pregnant, nursing, or interested in becoming pregnant within the next 3 years from the time of screening.
27. Participation as a subject in any other clinical studies involving medical devices or drugs in the last 30 days prior to surgery
28. A pending personal litigation relating to spinal injury (worker's compensation is not exclusionary).
29. Anticipated or potential relocation greater than 50 miles that may interfere with completion of follow-up examinations.
30. A mental illness or belongs to a vulnerable population, as determined by the investigator (e.g., prisoner or developmentally disabled), that would compromise ability to provide informed consent or compliance with follow-up requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with fusion success at the treated posterior anatomy of each level. | 12 months post procedure
  An individual subject is considered a fusion success if there is evidence of bridging trabecular bone across the posterior anatomy identified at both index levels determined using thin-slice CT and assessed by a third-party core imaging laboratory.
Proportion of participants with freedom from serious adverse event with definite relationship to treatment devices (interbody or posterior devices). | 12 months post procedure
  The seriousness and relationship of each adverse event will be adjudicated by a clinical events committee. A subject will be considered a primary endpoint failure if an adverse event is determined by the committee to be serious and to have a relationship to any of the devices used in the procedure including both interbody and posterior devices.
Proportion of Participants with freedom from injections (steroid, facet joint, nerve block) or subsequent revision surgery at index levels for symptoms related to back or leg pain. | 12 months post procedure
  A subject will be considered a primary endpoint failure if they require injections or subsequent revision surgery to treat new or recurrent symptoms of back or leg pain after their index surgery.

SECONDARY OUTCOMES:
Proportion of participants with the presence of Interbody bridging bone. | 12 month visit
  An individual subject is considered a success if there is evidence of bridging trabecular bone across the interbody space identified at both index levels determined using thin-slice CT and assessed by a third-party core imaging laboratory.
Differences in average segmental range of motion of the treated levels | 12 month visit
  Range of motion for each of the two treated levels will be measured by a third-party core imaging lab.
Differences in average change in disc height of the treated levels | 12 month visit
  Change in disc height for each of the two treated levels will be measured between the week-6 and 12-month visits by a third-party core imaging lab.
Proportion of participants with freedom from injections (steroid, facet joint, nerve block) or subsequent revision surgery at treated levels for symptoms related to back or leg pain. | through 24 month visit
  A subject will be considered a failure for this endpoint if they require injections or subsequent revision surgery to treat new or recurrent symptoms of back or leg pain after their index surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Summerside, PhD, Study Director — Providence Medical Technology

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD will be shared on a case-by-case basis after review of proposals by the Sponsor and Investigators.

REFERENCES:
- See also: Services US Department of Health and Human. Guidance document for the preparation of IDEs for spinal systems. Washington (DC): Food and Drug Administration Center for Devices and Radiological Health. 2000. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/guidance-document-preparation-ides-spinal-systems-guidance-industry-andor-fda-staff